CLINICAL TRIAL: NCT00410891
Title: Topical Antibiotics and Intravitreous Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Ta, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 96803 (eProtocol 4384)
Record Dates: First submitted 2006-10-02; First posted 2006-12-13 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Intravitreous; Injections
MeSH Terms: interventions — Gatifloxacin

ARMS (1):
- topical antibiotic (Experimental): topical gatifloxacin 4 times per day
  Interventions: Drug: gatifloxacin

INTERVENTIONS:
Drug: gatifloxacin

SUMMARY:
Evaluation of efficacy of topical preoperative antibiotics in patients undergoing intravitreous injections.

ELIGIBILITY:
Inclusion Criteria:

* intravitreous injection

Exclusion Criteria:

* antibiotic use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ta, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Antibiotic: topical gatifloxacin 4 times per day
  gatifloxacin
Period: Overall Study
Arm/Group | Topical Antibiotic
Started | 129
Completed | 129
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: patient undergoing IVT
Arm/Group | Topical Antibiotic
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 77 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 48
Conjunctival Bacterial Flora [Number; unit: percentage of patients] — Percentage of patients with bacterial isolates of interest in the eye prior to administration of study treatment
  percentage of patients
    Coagulase-negative staphylococcus | 75
    Staphylococcus aureus | 7
    Gram-negative rods | 6
    Streptococcus species | 7

OUTCOME MEASURES:

1. Primary Outcome: Positive Culture
Description: The percentage of patients with a positive bacterial culture following administration of study treatment is presented.
Time Frame: Study day 1, assessed following administration of study treatment
Measure: Number; unit: percentage of patients
Arm/Group | Topical Antibiotic
Number analyzed (Participants) | 129
percentage of patients | 8

ADVERSE EVENTS:
Time Frame: Study day 1 (average 1 hour)
Arm/Group | Topical Antibiotic
Serious Adverse Events (participants affected / at risk) | 0/129
Other Adverse Events (participants affected / at risk) | 0/129

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No